CLINICAL TRIAL: NCT02463500
Title: UT Southwestern Diabetic Foot Ulcers (DFU) and Osteomyelitis (DFO) Recruitment Database, Data and Tissue Repository
Acronym: DFUDatabase
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Larry Lavery, Professor, Department of Plastic Surgery, University of Texas Southwestern Medical Center
Other Study IDs: 18776
Record Dates: First submitted 2015-04-16; First posted 2015-06-04 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot Ulcers; Osteomyelitis
MeSH Terms: conditions — Diabetic Foot; Osteomyelitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood, bone and tissue samples will be banked in the UT Southwestern Department of Plastic Surgery Laboratory and tested for bacteria, biomarkers, inflammatory cytokines and other indicators of infection.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DFU with/without osteomyelitis: Patients of the investigators. Male and female, age 18 and older (up to age 89), of any race or ethnicities, who have diabetes (Type I or II) and a foot ulceration.
  Interventions: Other: DFU

INTERVENTIONS:
Other: DFU — Standard care.

SUMMARY:
This will be a continuing, prospective study of diabetic foot ulcers and infections, risk factors and clinical outcomes and a limited data set conducted by the investigator through the establishment of a data and tissue repository in the uT Southwestern Department of Plastic Surgery. in addition, subjects consented for this research will be asked about inclusion in a recruitment database to be used in the recruitment of subjects for future research on diabetic foot complications.

about 250 patients are seen for diabetic foot ulcers and infections each year.

DETAILED DESCRIPTION:
Subjects will be consented during a scheduled visit for standard care at the Clements University Hospital, UT Southwestern Wound Clinic, Parkland Hospital or the Parkland ASC Wound Clinic. There will be 2 study visits: Baseline and operating room visit. At the time of scheduled procedures or laboratory blood draws (as part of standard of care or SOC), soft tissue (from wound debridement or surgery), and bone if possible (from surgery or bone biopsy) will be obtained for histological sectioning and/or laboratory analysis. Tissue and or bone (surgical waste will be sent to the plastic surgery laboratory for storage and analysis.

Tissues with or without bone will be sent to the clinical pathology core for paraffin/frozen sectioning. Histological sections will be used for immunostaining and laser capture microdissection to evaluate tissue ultrastructure and region /cell specific gene expression analysis. Samples will also be sent to the Research and Testing Laboratory in Lubbock, TX for bacterial analysis and to Dermagenesis, LLC in Pompano Beach, FL for isolation of cellular components from different wound specimens and to define characteristics such as proliferation and migration rates. Bone (surgical waste) will also be sent to the 1st Department of Internal Medicine, Laiko General Hospital, Medical School, National and Kapodistrian University of Athens, Athens, Greece, for isolation of cellular components and cytokine analysis. In case infected bone is collected during surgery, it will be fixed and processed in the imaging core laboratory of our facility to evaluate biofilm with a Scanning Electron Microscope.

Relevant information obtained from the medical record will include age, gender, ethnicity, size (dimensions) of ulcer, location of ulcer, duration of ulcer, results of neurological and vascular testing, medical comorbidities, social history, laboratory data, offloading, and history of prior treatment (limited data set with no personal identifying information). Patient information will be de-identified and assigned a code. Bone and tissue samples will be banked in the UT Southwestern Department of Plastic Surgery Laboratory and tested for bacteria, biomarkers, inflammatory cytokines and other indicators of infection. All samples will be kept under the control of the principal investigator and used until exhausted. We will also follow these subjects for two (2) years to identify incidents of care and hospital readmissions for diabetic foot complications through review of the subject's electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

Patients of the investigators. Male and female, age 18 and older (up to age 89), of any race or ethnicities, who have diabetes (Type I or II) and a foot ulceration.-

Exclusion Criteria:

* Not meeting Inclusion Criteria.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the investigators. Male and female, age 18 and older (up to age 89), of any race or ethnicities, who have diabetes (Type I or II) and a foot ulceration.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2023-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 12 Weeks
  Wound healing defined as fully epithelialized over the base.
Biomarkers | 2 Years
  Quantity and types of biomarkers in blood, tissue and bone specimens
Adverse Events | 1 Years
  Number and type of adverse events, severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lavery, DPM, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas